CLINICAL TRIAL: NCT06835270
Title: Investigation of Different Treatment Approaches in Elderly Individuals With Chronic Nonspecific Low Back Pain: A Comparative Randomized Study
Brief Title: Investigation of Different Treatment Approaches in Elderly Individuals With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Kevser Gürsan, Principal Investigator, Uşak University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15/18
Record Dates: First submitted 2025-02-07; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Chronic Nonspecific Low Back Pain; Elderly (People Aged 65 or More)
Keywords: Yoga; electrotherapy; kinesiology taping; chronic nonspecific low back pain; elderly

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- The group that received standard physiotherapy approaches (Other): therapeutic ultrasound, hotpack and TENS (5x5 cm electrodes, applied to the thoracic 12 and sacral 1 regions).
  Interventions: Device: Standard physiotherapy approaches
- The group that received yoga interventions (Experimental): Yoga Group practiced Iyengar yoga asanas, pranayama, and mental focusing components in a group exercise format for 45 minutes.
  Interventions: Other: Yoga Exercises
- Kinesiology taping group (Experimental): In the kinesiology taping technique, tape was applied in an I-shape parallel to the m. quadratus lumborum muscle.
  Interventions: Other: Kinesiology taping
- The group that received educational sessions on low back pain (Other): The educational training was based on the WHO's guidelines for back pain.
  Interventions: Behavioral: Awareness training for low back pain

INTERVENTIONS:
Other: Yoga Exercises — Yoga group practiced Iyengar yoga asanas, pranayama, and mental focusing components in a group exercise format for 45 minutes.The yoga group was advised to practice yoga exercises at home following their yoga sessions.
  Arms: The group that received yoga interventions
Device: Standard physiotherapy approaches — Standard physiotherapy approaches group ( standard physiotherapy approaches (therapeutic ultrasound, hotpack) and TENS (5x5 cm electrodes, applied to the thoracic 12 and sacral 1 regions). Four electrodes were applied for 20 minutes with a pulse width of 50-100 µs and a frequency of 60-120 Hz. This group was additionally recommended to perform home exercises
  Arms: The group that received standard physiotherapy approaches
Other: Kinesiology taping — In the kinesiology taping technique, tape was applied in an I-shape parallel to the m. quadratus lumborum muscle. Interventions were conducted three times a week for four weeks, totaling 12 sessions.This group was additionally recommended to perform home exercises
  Arms: Kinesiology taping group
Behavioral: Awareness training for low back pain — The educational training was based on the WHO's guidelines for back pain. This group was additionally recommended to perform home exercises.
  Arms: The group that received educational sessions on low back pain

SUMMARY:
Chronic nonspecific low back pain (CNSLBP) is a common issue among the elderly, affecting their physical health, daily activities, sleep quality, and overall quality of life. This study aimed to compare the effects of various interventions, including standard therapy (ST), transcutaneous electrical nerve stimulation (TENS), yoga, kinesiology taping (KT), awareness education, and home exercises on pain, disability, sleep quality, and quality of life in elderly with CNSLBP. In line with the objectives of this randomized controlled trial, the following hypotheses have been formulated:

Hypothesis 1: Standard treatment and transcutaneous electrical nerve stimulation (TENS) have an effect on pain, disability status, sleep, and quality of life in elderly individuals with chronic non-specific low back pain (CNSLBP).

Hypothesis 2: Yoga has an effect on pain, disability status, sleep, and quality of life in elderly individuals with CNSLBP.

Hypothesis 3: Educational sessions and home exercise programs have an effect on pain, disability status, sleep, and quality of life in elderly individuals with CNSLBP.

Hypothesis 4: Kinesiology taping and home exercise programs have an effect on pain, disability status, sleep, and quality of life in elderly individuals with CNSLBP.

The study was conducted at a private physical therapy and rehabilitation center in the Aegean region between July 2024 and November 2024.

Patients were randomly assigned to four different groups. Group 1 (G1): Participants received standard physiotherapy approaches, including therapeutic ultrasound and hot packs, in addition to transcutaneous electrical nerve stimulation (TENS). TENS was applied using two channels with 5x5 cm electrodes placed over the thoracic 12 and sacral 1 regions. Four electrodes were used for 20 minutes with a pulse width of 50-100 µs and a frequency of 60-120 Hz.

Group 2 (G2): Participants engaged in Iyengar yoga sessions that included asanas, pranayama, and mental focus exercises. The sessions lasted 45 minutes and were conducted as group exercises tailored for elderly individuals. Additionally, participants were encouraged to continue yoga exercises on non-session days.

Group 3 (G3): Participants received educational sessions and home exercise programs targeting low back pain. The educational sessions were based on the World Health Organization (WHO) guidelines for low back pain management.

Group 4 (G4): Participants received kinesiology taping and home exercise programs. Kinesiology taping was applied in an I-shaped parallel manner to the quadratus lumborum muscle.

All interventions were administered three times per week for four weeks, totaling 12 sessions.

DETAILED DESCRIPTION:
With the rapid advancements in technology and medicine, life expectancy worldwide is steadily increasing, leading to a growing proportion of the elderly population. It is estimated that in the coming years, one in six individuals will be aged 60 or older. This demographic shift necessitates a more focused examination of health issues prevalent among older adults and the development of effective interventions.

The aging process is characterized by a progressive decline in cellular functions, resulting in adverse effects on physical health. One of the most prominent consequences of aging is musculoskeletal disorders. In particular, low back pain (LBP) is among the most prevalent conditions affecting elderly individuals and is directly associated with disability and a decline in quality of life. Notably, a substantial proportion of LBP cases occur without an identifiable underlying pathology and often become chronic, significantly impairing daily activities.

In the coming years, the prevalence of LBP is expected to rise considerably due to the aging population. This condition not only contributes to physical discomfort but also restricts mobility, increases dependency in daily activities, and negatively impacts sleep quality. The coexistence of chronic pain and sleep disturbances further exacerbates the decline in overall well-being among older adults. Consequently, identifying effective treatment strategies specifically targeting elderly individuals has become increasingly critical.

A variety of pharmacological and non-pharmacological approaches are available for managing LBP. However, pharmacological treatments may not always be the optimal solution, as they can pose risks of adverse effects, particularly in older adults. Non-pharmacological interventions, including yoga, electrotherapy, kinesiology taping, educational programs, and home-based exercise regimens, have been explored as alternative treatment modalities. Nevertheless, the existing body of research on these approaches remains limited, and further evidence is required, particularly concerning their efficacy in elderly populations.

This study aims to evaluate the effectiveness of different treatment modalities for elderly individuals suffering from chronic LBP. Various interventions, including standard physical therapy, electrotherapy, yoga, kinesiology taping, home exercise programs, and educational sessions, were compared to determine their effects on pain relief, mobility, sleep quality, and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Be able to understand verbal and visual communications
* Be literate
* To volunteer for the study
* Be 65 years of age or older
* Have Chronic Non-Specific Low Back Pain (CNSLBP)

Exclusion Criteria:

* Individuals who wish to withdraw from the study
* Those with spinal infections, radiculopathy, myelopathy, autoimmune diseases, spondylolysis, spondylolisthesis, spinal fractures
* Cardiovascular or pulmonary diseases that may contraindicate participation."

Ages: 65 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 63 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Pain Assesment | 4 weeks
  The Visual Analog Scale (VAS) is a commonly used tool in clinical settings to measure subjective characteristics or feelings that cannot be directly measured, such as pain intensity, fatigue, or mood. It typically consists of a straight line, often 10 cm in length, with two endpoints representing extreme levels of the phenomenon being measured.
  Ends of the scale: The left end (0) usually represents the absence of the characteristic (e.g., "No pain"), and the right end (10) represents the maximum intensity or severity of that characteristic (e.g., "Worst possible pain").
  Patient's response: The patient marks a point on the line that represents their perception of the current intensity. The position of the mark is then measured in millimeters or centimeters.Pain: The VAS might be used to assess pain, with one end of the line representing "No pain" and the other representing "Worst pain imaginable."
Disability Assessment | 4 weeks
  The Oswestry Disability Index (ODI) is a widely used clinical tool designed to measure the degree of disability in patients with low back pain. It assesses the impact of back pain on a person's daily activities, quality of life, and ability to function. The ODI is often used in both clinical practice and research to track changes in disability over time, particularly in individuals with chronic or acute low back pain.The ODI consists of 10 questions, each with 6 possible responses. Each question is related to a specific activity or aspect of life that could be impacted by low back pain. The responses are scored on a scale from 0 (no disability) to 5 (maximum disability), and each section is then given a score that reflects the severity of the disability.

SECONDARY OUTCOMES:
Sleep Quality Assesment | 4 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used self-reported questionnaire that assesses the quality and patterns of sleep over a 1-month period. It is designed to measure various aspects of sleep, including sleep duration, sleep disturbances, and overall sleep quality. The PSQI is useful for identifying sleep disorders and monitoring changes in sleep quality over time, especially in clinical and research settings.The PSQI consists of 19 questions that are grouped into 7 components. Each component is scored individually, and the sum of the scores determines the overall sleep quality. The seven components assess different aspects of sleep and its impact on daily life.
Quality of life assessment | 4 weeks
  The SF-36 (Short Form 36) is a widely used health survey tool designed to assess an individual's overall health status and quality of life. It is a generic, multidimensional measure of health that evaluates physical and mental well-being, and is often used in clinical practice, research, and health policy settings. The SF-36 is particularly useful for comparing the impact of different diseases, treatments, or interventions on individuals' health.
  The SF-36 consists of 36 items organized into 8 scales that measure various dimensions of health. These scales cover both physical and mental aspects of health, with questions on general health perceptions, functional status, and emotional well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Kevser Gursan, Dr., Principal Investigator — Uşak University
Locations (1):
- İzmir Private Rehabilitation Centre, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No